CLINICAL TRIAL: NCT04692610
Title: Effect of Prehabilitation on Stoma Self-Care, Anxiety, Depression and Quality of Life in Stoma Patients: A Randomized Controlled Trial
Brief Title: Effect of Stoma Prehabilitation on Stoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cihangir Akyol (Other)
Responsible Party: Sponsor-Investigator, Cihangir Akyol, Associate Proffessor, Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: U1111-1263-2558
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Stoma; Anxiety; Depression; Quality of Life
Keywords: Stoma; Self-care; prehabilitation; anxiety; depression; quality of life
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: 218 patients were included in the analysis.
  Each group had a different protocol:
  Group A - Postoperative Group received stoma education and stoma care after surgery beginning from the postoperative day-1; Group B - Pre- and Postoperative Group received stoma education both before surgery and on the postoperative day-1. They received stoma care postoperatively as usual; Group C - Prehabilitation Group received the same protocol as Group B, however in addition they were prehabilitated with a water-filled stoma pouch (250 ml) 48 hours before surgery (Figure 2). These pouches were not removed until surgery, and EST nurse preoperatively taught the patients how to manage the stoma pouch with similar standards as the usual postoperative stoma-care.
  The goal of the present study was to evaluate the stoma self-care ability, anxiety, depression and QoL of patients who underwent colorectal surgery and faecal diversion, and focusing on the effect of prehabilitation.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Placebo Comparator): Postoperative Education Group received stoma education and stoma care after surgery beginning from the postoperative day-1. In the preoperative period they were informed about stoma and stoma sites were marked.
  Interventions: Behavioral: postoperative stoma education; Behavioral: Postoperative stoma care
- Group B (Active Comparator): Pre- and Postoperative Education Group received stoma education both before surgery and on the postoperative day-1. They received stoma care postoperatively as usual. In the preoperative period they were also informed about stoma and stoma sites were marked.
  Interventions: Behavioral: preoperative stoma education; Behavioral: postoperative stoma education; Behavioral: Postoperative stoma care
- Group C (Experimental): Prehabilitation Group received the same protocol as Group B, however in addition they were prehabilitated with a water-filled stoma pouch (250 ml) 48 hours before surgery. These pouches were not removed until surgery, and EST nurse preoperatively taught the patients how to manage the stoma pouch with similar standards as the usual postoperative stoma-care.
  Interventions: Behavioral: Stoma prehabilitation; Behavioral: preoperative stoma education; Behavioral: postoperative stoma education; Behavioral: Postoperative stoma care

INTERVENTIONS:
Behavioral: Stoma prehabilitation — A stoma pouch was attached to the marked stoma site on the patient's abdominal surface after stoma education (only in group C). EST nurse filled 250 ml water into the pouch. Patients lived with these pouches until surgery. They experienced walking, sitting, sleeping, changing clothes with a pouch. They learned how to empty it. When a leak occurred, the pouch was changed by the nurse
  Arms: Group C
Behavioral: preoperative stoma education — A consultation period for stoma education by an EST nurse was approximately 45 minutes. Patients were shown pictures of a stoma. The stoma-care equipments and a pouch were also shown to the patients and they were informed about these equipments. They were also provided information about daily living with a stoma.
  Arms: Group B; Group C
Behavioral: postoperative stoma education — A consultation period for stoma education by an EST nurse was approximately 45 minutes. Patients were shown pictures of a stoma. The stoma-care equipments and a pouch were also shown to the patients and they were informed about these equipments. They were also provided information about daily living with a stoma.
Behavioral: Postoperative stoma care — Usual stoma care given by enterostomal therapy nurse after a surgery with fecal diversion

SUMMARY:
Stoma has serious psychosocial effects on patients. Stoma prehabilitation has a potential to overcome these problems. Patients in prehabilitation group were attached with a water-filled stoma pouch (250 ml) 48 hours before surgery. These pouches were not removed until surgery, and enterostomal therapy nurse preoperatively taught the patients how to manage the stoma pouch with similar standards as the usual postoperative stoma-care.

This study aims to measure the effects of prehabilitation on stoma self-care, quality of life, anxiety and depression levels.

DETAILED DESCRIPTION:
Stoma has serious psychosocial effects on patients. Stoma prehabilitation has a potential to overcome these problems. Patients in prehabilitation group were attached with a water-filled stoma pouch (250 ml) 48 hours before surgery. These pouches were not removed until surgery, and enterostomal therapy nurse preoperatively taught the patients how to manage the stoma pouch with similar standards as the usual postoperative stoma-care.

This study aims to measure the effects of prehabilitation on stoma self-care, quality of life, anxiety and depression levels.

A total of 240 patients met the inclusion criteria and were randomly assigned into three groups with the use of a prepared computerized block design by the biostatistician. Twenty-two patients were excluded and 218 patients were included in the analysis.

Each group had a different protocol:

Group A - Postoperative Group received stoma education and stoma care after surgery beginning from the postoperative day-1; Group B - Pre- and Postoperative Group received stoma education both before surgery and on the postoperative day-1. They received stoma care postoperatively as usual; Group C - Prehabilitation Group received the same protocol as Group B, however in addition they were prehabilitated with a water-filled stoma pouch (250 ml) 48 hours before surgery. These pouches were not removed until surgery, and enterostomal therapy (EST) nurse preoperatively taught the patients how to manage the stoma pouch with similar standards as the usual postoperative stoma-care.

Stoma site marking: Preoperative stoma site marking improves patients' QoL and independence in the postoperative period and decreases postoperative complications. In elective cases this should be considered as a must. In the current study all the patients' stoma sites were marked preoperatively by an EST nurse according to some important rules. Patients' abdominal surfaces were observed carefully for folds, scars, and creases in lying and standing positions. Bilateral points were chosen by paying attention to the planned incision line and the borders of the rectus muscle. At the end we had all the patients confirm they can see the marked sites.

Stoma education: A consultation period for stoma education by an EST nurse was approximately 45 minutes. Patients were shown pictures of a stoma. The stoma-care equipments and a pouch were also shown to the patients and they were informed about these equipments. They were also provided information about daily living with a stoma.

Stoma prehabilitation: A stoma pouch was attached to the marked stoma site on the patient's abdominal surface after stoma education (only in group C). EST nurse filled 250 ml water into the pouch. Patients lived with these pouches until surgery. They experienced walking, sitting, sleeping, changing clothes with a pouch. They learned how to empty it. When a leak occurred, the pouch was changed by the nurse.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent elective colorectal surgery and faecal diversion in the Ankara University Department of General Surgery between 2011 and 2016
* Patients with malignancy,
* Patients with polyposis syndrome,
* Patients with inflammatory bowel disease,
* Patients with diverticular disease
* Patients with perianal benign diseases

Exclusion Criteria:

* those who underwent emergency surgery
* those who developed stoma complications
* disoriented patients who could not cooperate
* patients with psychiatric disease
* patients with noncurable malign disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-11-15 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Stoma self-care ability | stoma follow-up was continued up to the 12th week
  All the patients with stoma were followed up by an enterostomal therapy nurse according to each group's own protocol. A stoma care follow-up form was completed beginning from the stoma education given by the nurse on the postoperative day-1 for all groups. Although patients in group C had learned how to manage a stoma pouch before surgery, their stoma-care follow-up forms were also completed after surgery beginning with the postoperative day-1. When the patient managed to empty the pouch with and without help, and when the patient was able to perform stoma care with the passive and active help of the nurse were recorded. And finally the day when the patient managed to perform stoma self-care was also recorded.

SECONDARY OUTCOMES:
Anxiety and depression score | postoperative 5th day
  Hospital anxiety and depression scale (HADS) has long been used to measure anxiety and depression, and has been validated for several times including Turkish population. According to the ROC analysis, the cut-off points of the Turkish form of the HAD scale were determined as 10 for the anxiety subscale and 7 for the depression subscale.
Stoma specific Quality of life | postoperative 4th week
  Quality of life was measured with the Stoma-QoL questionnaire which is an internationally recognized global feature. It has been validated in Turkish patients. The Stoma-QoL questionnaire covered 4 domains: sleep, sexual activity, relations to family and close friends, and social relations outside family and close friends. Each item uses a Likert scale from 1 to 4 and the total score ranges from 20 to 80.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet A Koç, MD, Principal Investigator — Ankara University School of Medicine Departmernt of General Surgery; Cihangir Akyol, MD, Study Chair — Ankara University School of Medicine Departmernt of General Surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koc MA, Akyol C, Gokmen D, Aydin D, Erkek AB, Kuzu MA. Effect of Prehabilitation on Stoma Self-Care, Anxiety, Depression, and Quality of Life in Patients With Stomas: A Randomized Controlled Trial. Dis Colon Rectum. 2023 Jan 1;66(1):138-147. doi: 10.1097/DCR.0000000000002275. Epub 2022 Feb 21. PMID 35195553